CLINICAL TRIAL: NCT06662734
Title: Infantile Versus Adult-type Fibrosarcoma and the Risk of Multiple Primary Malignancies: a Retrospective Cohort Based on SEER Database
Brief Title: Infantile Versus Adult-type Fibrosarcoma and the Risk of Multiple Primary Malignancies
Status: Completed | Type: Observational
Sponsor: asmaa salama ibrahim (Other)
Responsible Party: Sponsor-Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Organization: Suez Canal University (Other)
Other Study IDs: A274
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Fibrosarcoma
Keywords: infantile fibrosarcoma; Fibrosarcoma; SEER
MeSH Terms: conditions — Fibrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Fibrosarcoma is a malignant tumor originating from mesenchymal tissues and consists of fibroblasts with various types of collagen production. It represents 10% of musculoskeletal sarcomas and less than 5% of all primary bone tumors. It affects middle-aged patients with the most common location in the femur and 70% long tubular bones. Studies reported that fibrosarcoma patients tend to develop a subsequent primary malignancy, the analysis showed a higher risk of SPMs even a decade following the initial diagnosis of fibrosarcoma.

SPMs affect the long-term survival of patients with soft tissue tumors, and since there are no available studies analyzing the risk of second primary malignancies in different types of fibrosarcomas, especially the infantile and adult-type. Therefore, the purpose of this study was to assess the risk of second primary malignancies following primary fibrosarcoma diagnosis for a better understanding of the nature of this rare neoplasm. The investigators used the Surveillance, Epidemiology and End Results (SEER) database to extract the data and calculate the standardized incidence ratio as Observed/Expected and the Excess risk for second primary malignancies with 95% Confidence Interval. Significance was achieved at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with fibrosarcoma from 2000 to 2021.
* Sequence 0 or 1.
* Histological types:

Infantile fibrosarcoma, Fibromyxosarcoma, Periosteal fibrosarcoma, Facial fibrosarcoma, Dermatofibrosarcoma, Central odontogenic fibrosarcoma, Ameloblastic fibrosarcoma

Exclusion Criteria:

* Patients with unknown histology type

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 12,783 patients diagnosed with fibrosarcoma between 2000 and 2021.
Sampling Method: Probability Sample
Enrollment: 12783 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized incidence ratio and excess risk of developing multiple primary malignancies following fibrosarcoma diagnosis | from Jan, 2000 till Dec, 2021
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) and calculated the Excess absolute risk for Multiple primary malignancies for fibrosarcoma patients
The standardized incidence ratio and excess risk of developing second primary malignancies for different subtypes of fibrosarcoma | from Jan, 2000 till Dec, 2021

SECONDARY OUTCOMES:
The standardized incidence ratio and excess risk of multiple primary malignancies in fibrosarcoma patients across different racial groups | from Jan, 2000 till Dec, 2021
The standardized incidence ratio and excess risk of multiple primary malignancies in both males and females in fibrosarcoma patients | from Jan, 2000 till Dec, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided